CLINICAL TRIAL: NCT04385394
Title: Bright Light Therapy as Augmentation of Depressive Symptoms as Measured by Changes in Beck Depression Inventory, Hamilton Rating Scale for Depression and Outcome Questionnaire-45 on Acute Psychiatric Floor
Brief Title: Bright Light Therapy as Augmentation of Depressive Symptoms on Acute Psychiatric Floor
Acronym: BLT
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 1507582-1
Record Dates: First submitted 2019-12-23; First posted 2020-05-12 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to explore if Bright Light Therapy (BLT) as augmentation of depression treatment on an acute psychiatric floor is feasible, helps alleviate depressive symptoms, improve functioning, and decrease length of stay on the psychiatric floor.

DETAILED DESCRIPTION:
Background:

Bright light therapy is an evidence-based treatment for seasonal depression (SAD), recently there is evidence that it has some efficacy in nonseasonal major depressive disorder (MDD) when used together with antidepressants.

BLT works via the patient's eyes through

1. Melanopsin (Intrinsic Photo receptor ganglion Cells)
2. Suprachiasmatic Nucleus (SCN, master clock) which follows a rhythmic change
3. Serotonin

A number of studies showed seasonal changes in serotonergic parameters, including brain serotonin concentration and turnover. There were no research on using the BLT on the acute inpatient floor to augment the antidepressant treatment. Yet, there is a great need for such augmentation as for Selective Serotonin Reuptake Inhibitors (SSRI) to take full effect 4-6 weeks needed. Moreover, patients with depression often do not spend enough time on the direct sun light, which exacerbate and prolong their depressed mood. The augmentation with the BLT on the acute psychiatric floor will help the antidepressant work, expedite the recovery, and potentially shortens the length of stay in the hospital, which in turn will lead to an economic saving and faster return of the patient into the community and to the workforce.

Method:

This is an observational, case series study. All patients that meet exclusion criteria will have equal chance to receive BLT. We will administer the questionnaires before the BLT and at the end of treatment. Patient will continue to receive the pharmacological and therapeutic treatment on psychiatric floor as usual during the BLT. We will evaluate the changes in the questionnaires before and after BLT treatment, the length of stay on the unit. We will analyze the contributing factors such as age, gender, duration of depressive symptoms, other psychiatric and medical comorbidities, social factors (homelessness, social support, etc), current psychiatric medications.

Eligible patients will be invited to participate and consent will be obtain.

* The type of light we use is the "Sun Box Sun Square +"
* Emits about 10,000 lux of light and is wide enough to be used for more than 2 people.
* 186 watts
* Full spectrum 5000k white light (without the UV)
* It has an inbuilt spectrally transparent prismatic diffuser that blocks UV, that does not filter the quality of light and will not yellow.
* Minimal heat and no bulb flutter.
* Where: Bedroom / Common sitting area
* Reading/ Having breakfast/ Watching tv/Drawing
* Just after awakening within an hour early morning
* 30 mins/day
* Must have eyes open, but not looking into the light
* Staff will monitor while the patients are under the BLT

ELIGIBILITY:
Inclusion Criteria:

* depressive symptoms on BDI (score 14 and above - eligible for BLT) and/or
* depressive symptoms on HAMD-17 (score 8 and above)

Exclusion Criteria:

* no report of depressive symptoms; manic symptoms, acute psychosis, schizophrenia, schizoaffective disorder, impending Electro Convulsive Therapy (ECT), retinal risk factors, lupus, bright light sensitivity, glaucoma, cataracts, retinal detachment, retinopathy, patients on photosensitizing meds (tetracycline, sulfonamides, psoralens, and phenothiazine antipsychotics)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: inpatients reporting depressive symptoms that meet inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
depression scores | 7 days
  changes in depression scores, administered before light therapy and prior to discharge (corresponds to the last session of light therapy)
Functioning scores | 7 days
  symptoms distress, interpersonal functioning, social role

SECONDARY OUTCOMES:
length of stay | 7 days
  duration of stay on an inpatient unit in days

CONTACTS AND LOCATIONS:
Overall Officials: Luba Leontieva, MD, PhD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No